CLINICAL TRIAL: NCT03731169
Title: A Randomized Controlled Trial of the Effect of Cytochrome P450 2C19 Genotype-Specific Dosing Plus TDM vs. TDM Alone on Reaching Therapeutic Voriconazole Blood Levels
Brief Title: CYP2C19 Genotype-Specific Dosing Plus TDM on Reaching Therapeutic Voriconazole Blood Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Marisa Battistella, Pharmacy Clinician Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-9226
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Aspergillosis Invasive; Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TDM Only (Active Comparator): This is the standard of care trial arm. Patients receive voriconazole dosages according to the product monograph. After day 4, dosing in both trial arms will adhere to the following in order to reach the target therapeutic window: 1.0-5.5 mg/L.
  Interventions: Drug: Standard of Care
- Genotyping + TDM (Experimental): After ascertaining CYP2C19 genetic status, the participants will be categorized as having either the ultra-rapid metabolizer (URM), extensive metabolizer (EM), heterozygous extensive metabolizer (HEM) or poor metabolizer (PM) phenotype. They will receive an experimental dosage regimen based on their phenotype. receive the following dosing regimen until TDM is conducted on day 4. After day 4, dosing in both trial arms will adhere to the following in order to reach the target therapeutic window: 1.0-5.5 mg/L.
  Interventions: Genetic: Voriconazole genotype-specific dosing

INTERVENTIONS:
Genetic: Voriconazole genotype-specific dosing — Those in the intervention arm will receive an experimental dosage regimen of voriconazole based on their genetic status.
  URM: 6 mg/kg voriconazole twice on the first day followed by 5 mg/kg twice daily, rounded to the nearest 50mg for oral formulations up to day 4 post-start of voriconazole therapy.
  EM: 6 mg/kg voriconazole twice on the first day followed by 4 mg/kg twice daily, rounded to the nearest 50mg for oral formulations up to day 4 post-start of voriconazole therapy.
  HEM and PM: 6 mg/kg voriconazole twice on the first day followed by 2 mg/kg twice daily, rounded to the nearest 50mg for oral formulations up to day 4 post-start of voriconazole therapy.
  Other Names: Genotype-guided dosing
  Arms: Genotyping + TDM
Drug: Standard of Care — Participants are given 6 mg/kg voriconazole twice on the first day followed by 4 mg/kg twice daily, rounded to the nearest 50mg for oral formulations up to day 4 post-start of voriconazole therapy. After TDM is conducted on day 4 for all patients, dosing in both trial arms will adhere to the following in order to reach the target therapeutic window: 1.0-5.5 mg/L.
  Arms: TDM Only

SUMMARY:
Invasive aspergillosis is a fungal infection which left untreated, is a significant cause of morbidity and mortality. Immunocompromised patient populations such as solid organ transplant and malignant hematology patients are especially susceptible to invasive fungal infections. Voriconazole is an anti-fungal agent that is frontline therapy for invasive aspergillosis. Treatment success is highly dependent on maintaining therapeutic voriconazole concentrations. The current published literature has established that treatment failure is associated with sub- and supra-therapeutic voriconazole concentrations.

Maintaining therapeutic voriconazole concentrations however, is challenging due to the high inter and intra-patient variability in voriconazole pharmacokinetics. The complex kinetics of voriconazole renders current manufacturers' dosing guidelines ineffective. Much of this complexity has been linked to genetic polymorphisms in the cytochrome P450 2C19 gene, and it has been found that CYP2C19 genotype plays an important role in determining voriconazole exposure levels. Therapeutic drug monitoring has been found to increase efficacy of voriconazole treatment through the monitoring of patients' voriconazole levels, allowing for dosage adjustments in response to supra- or sub-therapeutic levels.

There are few robust studies that have examined the effect of CYP2C19 genotype on voriconazole treatment outcomes. They have been unable to determine relationships between CYP2C19 genetic status, and clinical efficacy and safety. No studies to our knowledge have made dosing adjustments based on CYP2C19 genetic status.

The study aim is to explore the utility of voriconazole dosing that is based on the genetic status of the patient in conjunction with therapeutic drug monitoring. Over the course of one year, solid organ transplant recipients at Toronto General Hospital and malignant hematology patients at Princess Margaret Cancer Centre receiving voriconazole therapy will be randomized into one of two trial arms: a control arm receiving therapeutic drug monitoring only, or a treatment arm receiving genotype-specific dosing in conjunction with therapeutic drug monitoring. The investigators will compare the proportion of patients that achieve voriconazole therapeutic concentrations, the number of dose adjustments needed to achieve therapeutic voriconazole levels, and clinical outcomes between trial arms.

DETAILED DESCRIPTION:
Purpose of Research:

Invasive aspergillosis (IA) is a fungal infection which left untreated, can cause dangerous complications and death. Transplant patients who have weakened immune systems are at higher risk of getting IA. Voriconazole is a medication that is prescribed for IA. In order for voriconazole to work, it is important to maintain the right amount of drug in the blood. The investigators check for the right amount of voriconazole in the blood by collecting blood samples. This process is called therapeutic drug monitoring (TDM) and usually done for transplant patients with weakened immune systems. However, maintaining the right amount of drug in the blood is still difficult since voriconazole is absorbed and excreted by the body differently for each person, depending on their genetic make-up. This study will try to understand if genetic testing early on in addition with TDM will be able to provide us with doses tailored to each individual.

Study Design:

Patients who consent to participate in this study and who are receiving voriconazole therapy for IA will be randomly split into one of two groups. The control group will receive voriconazole dosages and then TDM according to the usual treatment for the patient's condition. A treatment group will receive altered dosages that are specific to their genetic make-up for the first four days of treatment and will then receive routine TDM. This altered dosing for the treatment group is experimental and is not routinely used in patients' care. TDM will take place at approximately the fourth day after starting voriconazole for all patients, and from this point on the usual treatment will resume for all patients.

Participation in the study will be for the entire amount of time the patient is taking voriconazole. The study staff will meet with the patient once, provided they meet the study criteria. This will be the only visit from the study staff. This visit will take place immediately after being prescribed voriconazole and is estimated to take 1-2 hours.

Should the patient decide to participate in the study, basic demographic information will be collected at this time and the patient's medical records will be accessible to the study staff. One saliva sample will be collected from the patient at this time for the genetic testing portion of the study. The genetic testing used in this study will be specific to looking at the way the patient's body handles voriconazole and will not inform us of any other potential condition. No incidental findings will be discovered. This procedure will be done by Spartan Bioscience, a third party company. The patient's saliva sample will be sent with a code and will not show the patient's name or address, or any information that directly identifies them. The patient's saliva sample will be immediately destroyed after the genetic testing component has been completed. The patient's genetic information will remain confidential as no research data will be shared with Spartan Bioscience or anyone outside the study staff. No additional procedures outside of routine care will be done. As part of routine care, the patient's treatment will be regularly be assessed by a physician.

ELIGIBILITY:
Inclusion Criteria:

* All adult malignant hematology patients who are prescribed voriconazole.

Exclusion Criteria:

* Patients that have previously taken voriconazole within the last 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Voriconazole trough concentrations at steady-state | 1 year
  To determine if the proportion of patients who achieve therapeutic voriconazole trough concentrations at steady-state through genotype-specific dosing in conjunction with TDM is greater than the proportion of patients who obtain therapeutic voriconazole concentrations via TDM alone.
Number of dose adjustments | 1 year
  To determine if genotype-specific dosing in conjunction with TDM will result in a fewer number of dose adjustments needed to achieve therapeutic voriconazole levels, compared to TDM alone.
Genotype-specific dosages | 1 year
  To evaluate the genotype-specific dosages suggested for the genotyping plus TDM trial arm.

SECONDARY OUTCOMES:
Genotype-specific dosing on treatment success/failure | 1 year
  To determine if genotyping can increase treatment success (complete or partial response), predict the incidence of voriconazole dose-related adverse events (AEs), severity of toxicity, and incidence of termination of voriconazole therapy due to voriconazole dose-related AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Battistella, PharmD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Cancer Care Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers.